CLINICAL TRIAL: NCT02242656
Title: A Phase 3, Open Label Responder Treatment Period With a Randomized, Blinded, Three-Period Crossover, Followed by an Open Label Safety Period to Evaluate the Clinical Efficacy, Safety, and Pharmacokinetics of Investigational Drug MP-101 (Opium Tincture and Opium Tincture With Reduced Uncharacterized Material) to Treat Chronic Diarrhea in Subjects With Short Bowel Syndrome Who Have Had an Inadequate Response to Anti-Diarrheals
Brief Title: A Phase III Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Investigational Product MP-101 in Subjects With Short Bowel Syndrome Who Have Had an Inadequate Response to Anti-Diarrheals
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Transfer of IND to new marketing authorization holder
Sponsor: Marathon Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-101-CL-001
Record Dates: First submitted 2014-09-10; First posted 2014-09-17 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-10

CONDITIONS: Short Bowel Syndrome; Short Gut Syndrome; SBS; Short Bowel; Short Gut
Keywords: Short Bowel Syndrome; SBS; Chronic Diarrhea; Short Bowel; Short Gut; Short Gut Syndrome; Anti-Diarrheal; Opium Tincture; loperamide; diphenoxylate; ileostomies; tincture of opium; DTO; codeine; morphine; opiate
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Assigned to receive Treatment A (Period 1), Treatment B (Period 2), Treatment C (Period 3)
  Interventions: Drug: Opium Tincture USP Deodorized
- Group 2 (Experimental): Assigned to receive Treatment B (Period 1), Treatment A (Period 2), Treatment C (Period 3)
  Interventions: Drug: Opium Tincture USP Deodorized

INTERVENTIONS:
Drug: Opium Tincture USP Deodorized — Treatment A - 0.6 mL, MP-101 (10 mg/mL, Opium Tincture (OT)), USP (Deodorized) QID oral drops, followed by Treatment B - 0.6 mL, MP-101, 1/12 dilution, (0.833 mg/mL, OT), USP (Deodorized) QID oral drops, followed by Treatment C - 0.6 mL, MP-101 (10 mg/mL Opium Tincture with reduced uncharacterized material) QID oral drops
  Arms: Group 1
Drug: Opium Tincture USP Deodorized — Treatment B - 0.6 mL, MP-101, 1/12 dilution, (0.833 mg/mL, OT), USP (Deodorized) QID oral drops, followed by Treatment A - 0.6 mL, MP-101 (10 mg/mL, Opium Tincture (OT)), USP (Deodorized) QID oral drops, followed by Treatment C - 0.6 mL, MP-101 (10 mg/mL Opium Tincture with reduced uncharacterized material) QID oral drops
  Arms: Group 2

SUMMARY:
MP-101 will be evaluated in this study to see if it is safe, tolerable, and can help people with Short Bowel Syndrome. This study will also find out if taking MP-101 can improve the symptoms of Short Bowel Syndrome and reduce the number of times subjects experience bowel movements.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female adults, 18 years of age or older at the time of consent
2. Have SBS that is inadequately controlled on current antidiarrheal medication (e.g., loperamide or diphenoxylate), including subjects with ileostomies, based on the 7 days prior to Day 1 of the study

   a. Subjects must be >3months post intestinal resection
3. Have a history of persistent loose stools for more than 4 weeks
4. Be on a combination of Opium Tincture and an anti-diarrheal (loperamide or diphenoxylate) or an anti-diarrheal agent alone
5. If currently taking Opium Tincture, be willing to stop the continued use of Opium Tincture at screening visit until the start of study treatment and willing to stop the use of any other anti-diarrheal for the duration of the study
6. Be able to maintain their current diet for the duration of the study
7. Be on stable nutritional support (parenteral or oral)
8. Males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months of natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy)
9. Females of childbearing potential must agree to use 1 of the following acceptable birth control methods:

   1. Surgically sterile (hysterectomy or bilateral oophorectomy)
   2. Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation)
   3. Intrauterine device (IUD) in place for at least 3 months
   4. Abstinence (not having sexual intercourse)
   5. Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening and through study completion
   6. Stable hormonal contraceptive for at least 3 months prior to study and through study completion
   7. Vasectomized partner
10. Females of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at screening
11. Be able to understand and provide signed informed consent

Exclusion Criteria:

1. Unable or unwilling to stop the use of Opium Tincture or any anti-diarrheal medication at the screening visit.
2. Have any history of or active neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease that is considered clinically significant, is not currently controlled by medication, and is stable as deemed by the Investigator
3. Have clinically significant electrocardiogram (ECG) abnormalities as determined by the PI or vital sign abnormalities (systolic blood pressure < 90 mmHg, diastolic blood pressure < 60 mmHg, or heart rate >100 bpm) at screening
4. Have clinically significant elevation of liver enzymes (> 3 times the upper limit of normal) or clinically relevant renal disease, (creatinine >1.5) or any other clinically significant abnormal laboratory test results found during medical screening as determined by the Principal Investigator
5. Have a history of major mental illness that in the opinion of the Investigator may affect the ability of the subject to safely participate and reliably complete the study
6. Have a history of alcohol or substance abuse within the past 2 years. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz. beer, 5.0 oz. wine, or 1.5 oz. distilled spirits)
7. Have a known allergy or intolerance to Opium Tincture or any of the excipients in the formulation (alcohol, opium, or morphine)
8. Is currently taking an opioid derivative (other than Opium Tincture) or any other medication which, in the opinion of the investigator, could interfere with the interpretation of the study results
9. Are currently taking antibiotics for bacterial overgrowth
10. Have participated in another interventional clinical trial within 30 days prior to screening with the exception of observational cohort studies or non-interventional studies.
11. Have known or suspected pregnancy, planned pregnancy, or lactation
12. Have a planned surgery over the course of the study
13. Have a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of responders between Treatments A and B for the Intent-To-Treat (ITT) population | Last day of Periods 1 (Days 16-17) and 2 (Days 25-26)
  30% or greater reduction in 24-hour stool volume from baseline

SECONDARY OUTCOMES:
Percentage of responders between Treatments A and B for the Modified-Intent-To-Treat (mITT) population | Last day of Periods 1 (Days 16-17) and 2 (Days 25-26)
  30% or greater reduction in 24-hour stool volume from baseline for subjects who complete both periods 1 and 2 of the randomized, blinded, crossover portion of the study
Establish non-inferiority of the percentage of responders between Treatment A and Treatment C | Last day of Period 3 (Day 34-35)
  30% or greater reduction in stool volume from baseline between Treatment A (with uncharacterized material) and Treatment C (with reduced uncharacterized material) for ITT and mITT efficacy population (subjects from the ITT population who complete both Treatments A and C)
24-hour stool volume comparison between Treatment A and B for ITT and mITT | Last day of Periods 1 (Day 16-17) and 2 (Day 25-26)
  Comparison of stool volume measurements
24-hour fecal events between Treatment A and B for ITT and mITT | Period 1 (Day 10-16) and 2 (Day 19-25)
  Changes in the number of 24-hour fecal events for ITT and mITT
24-hour nocturnal fecal events between Treatment A and B for ITT and mITT | Period 1 (Day 10-16) and 2 (Day 19-25)
  Changes in the number of 24-hour nocturnal (ad defined for each subject) fecal events for ITT and mITT
Single and multiple dose Pharmacokinetic (PK) parameters | Day-1, Day 1, Day 7, Day 57-59
  Evaluate the pharmacokinetics of morphine, codeine, thebaine and papaverine after single dose and multiple dose administration of MP-101
Number of Participants with Adverse Events | Up to 60 Days
  Review of safety events throughout the course of the study
Number of Participants Up-Titrated | Days 35-60
  Review of safety events throughout the course of the study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Cleveland Clinic, Cleveland, Ohio
  - Regional Infectious Diseases Infusion Center, Lima, Ohio
  - Vanderbilt Center for Human Nutrition, Nashville, Tennessee